CLINICAL TRIAL: NCT00189514
Title: Extension Study of Protocol 137OB-201 to Examine the Long Term Effect of Pramlintide on Body Weight and Its Safety and Tolerability in Obese Subjects
Brief Title: A Study to Examine the Long Term Effect of Pramlintide on Body Weight and Its Safety and Tolerability in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 137OB-201E
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: obesity; weight loss; Amylin; pramlintide
MeSH Terms: conditions — Obesity; Weight Loss | interventions — pramlintide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: pramlintide acetate
- 2 (Experimental)
  Interventions: Drug: pramlintide acetate
- 3 (Experimental)
  Interventions: Drug: pramlintide acetate
- 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pramlintide acetate — Subcutaneous injection, twice a day or three times a day, at doses of 120mcg, 240mcg, or 360mcg
  Other Names: Symlin
  Arms: 1; 2; 3
Drug: placebo — subcutaneous injection, three times a day, volumes equivalent to 120mcg, 240mcg, or 360mcg of pramlintide acetate
  Arms: 4

SUMMARY:
This is a long term extension to study 137OB-201 which is designed to examine the effect of pramlintide on body weight and its safety and tolerability in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed Protocol 137OB-201.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Examine the long-term effect of subcutaneously (SC) injected pramlintide on body weight in obese subjects. | open ended
Examine the long-term safety and tolerability of SC injected pramlintide in obese subjects. | open ended

SECONDARY OUTCOMES:
Investigate the long-term effect of SC injected pramlintide in obese subjects on various anthropometric and pharmacodynamic parameters. | open ended

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (21):
- United States (21):
  - Research Site, Chula Vista, California
  - Research Site, San Diego, California
  - Research Site, Walnut Creek, California
  - Research Site, Miami, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Olympia, Washington

REFERENCES:
- [Derived] Smith SR, Aronne LJ, Burns CM, Kesty NC, Halseth AE, Weyer C. Sustained weight loss following 12-month pramlintide treatment as an adjunct to lifestyle intervention in obesity. Diabetes Care. 2008 Sep;31(9):1816-23. doi: 10.2337/dc08-0029. Epub 2008 Jun 20. PMID 18753666